CLINICAL TRIAL: NCT05405322
Title: Inclusive Programme for the Optimisation of Health and Well-being of HIV-positive Young People (15-24 Years) and for the Promotion of Their Community Representation in Senegal and Burkina Faso (2021 => 36 Months) (TRANSITIONS)
Brief Title: Improving Care and Community Representation for Adolescents and Young Adults Living With HIV in West Africa
Acronym: TRANSITIONS
Status: Active, not recruiting | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Sidaction (Other); EXPERTISE FRANCE, Paris France (Unknown); Children and HIV Network in AFRICA (EVA), Dakar Senegal (Unknown); Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Principal Investigator, Cecile Cames, Dr, Institut de Recherche pour le Developpement
Other Study IDs: 999999
Record Dates: First submitted 2021-11-10; First posted 2022-06-06 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Adolescent Behavior; Transition
Keywords: adolescent; HIV infection; transition; west africa; community; peer
MeSH Terms: conditions — HIV Infections; Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Context: HIV-positive young people aged 15 to 24 are a heterogeneous population in terms of gender, age, mode of transmission, sexual orientation and risk-taking. This most vulnerable age group is at greater risk of disruption of medical care and poor compliance, and has greater needs for psychosocial support and differentiated health services. It remains highly invisible in West African countries, both in the definition of care policies and in the allocation of resources and community representation.

Objectives: The overall objective of the project is to contribute to the improvement of retention in care, health and well-being of adolescents and young adults living with HIV (AYAHIV) and to support their integration into the community space.

SO1: Support the operationalisation of the transition of HIV-infected adolescents from paediatrics to adult medical services in a stakeholder inclusive, participatory and responsive approach SO2: Contribute to the empowerment and autonomy of adolescents and young adults living with HIV in the project environment SO3: Contribute to the generation and dissemination of evidence-based information and recommendations on the situation and needs of adolescents and young adults, including key populations, living with HIV

Target: Approximately 67 caregivers∙e∙s ≥ 25 years old, of which 64%F, 30 peer-referent associations of 20-24 years old (ratio F/H= 1:1), 700 AYAHIV ≥ 15 years old, of which 47%F, in paediatrics and 500-600 AYAHIV aged 15-24 years old in adult medicine, of which 41%F, and including AYAHIV associations Summary of activities: Based on the capitalisation and pooling of experiences of partner teams, the project proposes to support the implementation of transition in a pragmatic approach, adapted to the needs of adolescents and inclusive of carers, adolescents and community peers. More globally, it contributes to improving the health, empowerment and autonomy of HIV-positive youth, including key populations, in particular through support to training, structuring and community representation of youth associations, documentation of the conditions of entry into care and their specific needs, including digital health, production and availability of evidence and recommendations in this West African context and advocacy building.

A multidisciplinary and participatory research-action project, carried out by the IRD in Senegal and financed by Sidaction, accompanies the three specific objectives of the project.

DETAILED DESCRIPTION:
Context: HIV-positive young people aged 15 to 24 are a heterogeneous population in terms of gender, age, mode of transmission, sexual orientation and risk-taking. This most vulnerable age group is at greater risk of disruption of medical care and poor compliance, and has greater needs for psychosocial support and differentiated health services. It remains highly invisible in West African countries, both in the definition of care policies and in the allocation of resources and community representation.

Objectives: The overall objective of the project is to contribute to the improvement of retention in care, health and well-being of adolescents and young adults living with HIV (AYAHIV) and to support their integration into the community space.

SO1: Support the operationalisation of the transition of HIV-infected adolescents from paediatrics to adult medical services in a stakeholder inclusive, participatory and responsive approach SO2: Contribute to the empowerment and autonomy of adolescents and young adults living with HIV in the project environment SO3: Contribute to the generation and dissemination of evidence-based information and recommendations on the situation and needs of adolescents and young adults, including key populations, living with HIV

Target: Approximately 67 caregivers∙e∙s ≥ 25 years old, of which 64%F, 30 peer-referent associations of 20-24 years old (ratio F/H= 1:1), 700 AYAHIV ≥ 15 years old, of which 47%F, in paediatrics and 500-600 AYAHIV aged 15-24 years old in adult medicine, of which 41%F, and including AYAHIV associations Summary of activities: Based on the capitalisation and pooling of experiences of partner teams, the project proposes to support the implementation of transition in a pragmatic approach, adapted to the needs of adolescents and inclusive of carers, adolescents and community peers. More globally, it contributes to improving the health, empowerment and autonomy of HIV-positive youth, including key populations, in particular through support to training, structuring and community representation of youth associations, documentation of the conditions of entry into care and their specific needs, including digital health, production and availability of evidence and recommendations in this West African context and advocacy building.

A multidisciplinary and participatory research-action project, carried out by the IRD in Senegal and financed by Sidaction, accompanies the three specific objectives of the project.

Expected impact :

* Seamless operationalisation of the supported and coordinated transition in care process and scaling up to the level of the 12 countries of the EVA network.
* Young associative actors are able to advocate to guide decision-makers, based on the evidence they have helped to produce (participatory approach)
* The ultimate change, expected at the end of the project, is that institutional stakeholders will integrate these recommendations into the national programme for the care of PLHIV, both operationally and financially.

ELIGIBILITY:
Inclusion Criteria:

* being HIV-infected
* aged 15 to 24 years
* on antiretroviral treatment
* HIV status disclosed
* caretaker's written consent (if < 18 years)
* adolescent's written consent

Exclusion Criteria:

* mental illness

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The target population of the study is all HIV-infected adolescents (mainly through mother-to-child transmission) aged 15 to 24 years, eligible for transition to care and followed up in the active files of reference centers that are members of the EVA network in Senegal and Burkina Faso.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
retention in care | Month 12
  percent of adolescents who remain in care
retention in care | Month 21
  percent of adolescents who remain in care

SECONDARY OUTCOMES:
virologic suppression | Month 12
  percent of adolescents who maintain or reach undetectable viral load
virologic suppression | Month 21
  percent of adolescents who maintain or reach undetectable viral load
quality of life in relation to health | Month 12
  percent of adolescents who improve their score of quality of life in relation to health
quality of life in relation to health | Month 21
  percent of adolescents who improve their score of quality of life in relation to health
level of preparedness to adult care | Month 12
  percent of adolescents who improve their score of preparedness to adult care

CONTACTS AND LOCATIONS:
Locations (4):
- Burkina Faso (2):
  - CHU CDG, Ouagadougou
  - CHU YO, Ouagadougou
- Senegal (2):
  - Chnear Albert Royer, Dakar
  - Centre hospitalier Roi Baudouin, Guédiawaye

REFERENCES:
- Available data/document: podcasts — https://www.ird.fr/positifs-une-collection-de-podcasts-pour-un-nouveau-regard-sur-les-jeunes-vivant-avec-le-vih-en — Experiences of participatoy research with the participants included in the Transitions Study and their peers.